CLINICAL TRIAL: NCT02314988
Title: Topical Application of Tranexamic Acid (CYKLOKAPRON®) to Reduce Blood Loss During Spine Surgery
Brief Title: Tranexamic Acid to Reduce Blood Loss in Spine Surgery
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ronald A. Lehman, Professor of Orthopaedic Surgery, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAQ6795; 201409111 (Other: Washington University)
Record Dates: First submitted 2014-12-03; First posted 2014-12-11 (Estimated); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Spinal Injuries; Spinal Deformity
Keywords: Tranexamic acid; Antifibrinolytic; Perioperative blood loss; Postoperative drain output; Allogenic transfusion
MeSH Terms: conditions — Spinal Injuries | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Subjects will receive tranexamic acid on the surgical wound.
  Interventions: Drug: Tranexamic Acid
- Placebo control (Placebo Comparator): Subjects will receive placebo (saline solution) on the surgical wound.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — 3.0 grams of tranexamic acid will be poured in the surgical field and left in contact for five minutes. Subsequently, excess study solution will be suctioned away without touching the surrounding tissue surfaces and then the would closed without irrigation or manipulation.
  TXA solution will be prepared using a dose of 3 grams of tranexamic acid combined with 70 mL of sterile normal saline, for a total volume of 100 mL.
  Other Names: Cyclokapron; TXA
  Arms: Intervention
Drug: Placebo — Placebo will be poured in the surgical field and left in contact for five minutes. Subsequently, excess solution will be suctioned away without touching the surrounding tissue surfaces and then the would closed without irrigation or manipulation.
  The placebo solution will be 100 mL of sterile normal saline.
  Other Names: Saline Solution
  Arms: Placebo control

SUMMARY:
This study is designed to evaluate the efficacy of topical tranexamic acid to reduce perioperative blood loss, reduction in postoperative drain output and allogenic transfusion requirements.

The proposed study will be a prospective, randomized, double-blind (subject, surgeons, investigators, research coordinators) placebo-controlled study. Patients requiring posterior spinal fusion will be enrolled for this study. Furthermore, patients undergoing elective complex deformity surgery will also be enrolled. Both populations of patients will be randomized into two groups. Group I will receive standard of care operative fixation with topical tranexamic acid intervention (test); Group II will receive standard of care operative fixation with normal saline (placebo) intervention. This study will have a 2-year follow-up and will consist of three periods: screening/enrollment phase up to 21 days from the day of injury to the day of randomization and operative intervention, an inpatient data collection period for 4 days postoperative, and then a follow-up period for 2-years postoperative (visits occurring at 16 weeks, 1 year, and 2 year) time points.

DETAILED DESCRIPTION:
Reducing perioperative blood loss is critically important in the treatment of multiply injured combat casualties, and major blood loss during complex spine trauma surgery is a significant concern. Similar to previous studies in dental, cardiac, and total knee arthroplasty procedures, the use of topical tranexamic acid during complex combat related spine trauma surgery can be a cost-effective and simple route of administration to reduce blood loss, with no significant systemic effects. Patients would be expected to benefit immediately by decreasing blood loss and the need for blood transfusion postoperatively, thereby exposing them to less risk of transfusion reactions or disease transmission. This may also potentially decrease the rate of surgical site infection because patients have been found to have a significantly increased risk for surgical site infection after blood transfusion due to changes in the immune system, and by also decreasing the amount of blood that collects under the surgical wound, which serves as excellent medium for bacterial growth. The goal of the investigators study is to determine if the use of topical tranexamic acid (TXA) in the setting of complex spine surgery reduces blood loss, and subsequently reduces the rate of allogenic blood transfusion and surgical site infection.

ELIGIBILITY:
Inclusion Criteria:

1. Thoracic or lumbar spinal column injury with or without neurologic deficit requiring surgical fixation
2. Surgical fixation to be performed within 21 days of injury
3. Adult patients undergoing long segment (>5 fusion levels) posterior spinal fusions

Exclusion Criteria:

1. Age <18 or >80 years old
2. Severe soft tissue disruption around planned surgical site preventing adequate primary wound closure
3. Physiologic instability or ongoing sepsis/infection
4. Use of intravenous tranexamic acid during the pre-study period
5. Ballistic spinal column injury
6. Allergy to tranexamic acid
7. Disturbances of color vision or color blindness
8. Pre-operative hemoglobin value of <7 g/dL, or <10 g/dL if patient has comorbidities or symptoms which will require pre-operative allogeneic blood transfusion
9. Refusal to consent for blood products
10. Participation in another clinical trial
11. Moderate or severe traumatic brain injuries that do not allow participation in individual patient outcomes surveys
12. Subarachnoid hemorrhage, anecdotal experience indicates that cerebral edema and cerebral infarction may be caused by TXA
13. Concomitant use of Factor IX Complex concentrates or Anti-inhibitor Coagulant concentrates, as the risk of thrombosis may be increased
14. Preoperative use of anticoagulant therapy (heparin, low-molecular weight heparin, warfarin) within three days before surgery, or non-steroid inflammatory medication (aspirin, ibuprofen, naprosyn) use within seven days before surgery
15. Fibrinolytic disorders requiring intraoperative antifibrinolytic treatment
16. Disseminated intravascular coagulation (DIC)
17. Coagulopathy (as identified by a preoperative platelet count of <150,000/mm3, an international normalized ratio of >1.4, or a prolonged partial thromboplastin time >1.4 times normal)
18. History of arterial or venous thromboembolic disease (such as a cerebrovascular accident, deep-vein thrombosis, or pulmonary embolus), as these patients may be at increased risk for venous or arterial thrombosis
19. Upper urinary tract or ureteral injury (ureteral obstruction due to clot formation in patients with upper urinary tract bleeding has been reported)
20. Pregnancy or breastfeeding (Category B)
21. Substantial renal dysfunction (as assessed by a serum creatinine > 1.5 or calculated creatinine clearance of < 50) or hepatic failure
22. Major co-morbidities: alcohol or drug abuse, illnesses that affect bone or calcium metabolism, connective tissue disorders, coronary artery disease, severe ischemic heart disease [New York Heart Association Class III or IV], previous myocardial infarction, severe pulmonary disease [forced expiratory volume <50% of normal], diabetes mellitus (Type I or Type II), immunosuppression, peripheral vascular disease, severe penetrating or hemorrhagic traumatic brain injury, a history of skeletal malignancies, prior external beam or implant radiation therapy involving the skeleton.
23. History of seizure or convulsive disorders, or currently concomitant use of other medications that are known to reduce seizure threshold
24. History of dural tear or open subdural space

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Maximal drop in systemic hemoglobin concentration during the postoperative period | Patients will be followed through postoperative day 4

SECONDARY OUTCOMES:
Reduction in the rate of surgical site infections | Duration of the hospital stay (an average of 2 weeks), first postoperative wound check visit
  Defined by decreasing the allogenic transfusion rate (an independent risk factor for surgical site infections) as well as by decreasing the formation of postoperative hematoma (a nidus for infection).
Number of complications | Up to postoperative day 4
  Defined as thromboembolic event, including deep vein thrombosis (DVT) or pulmonary embolism (PE)
Systemic absorption of locally applied drug | Baseline (pre-surgery), immediately after administration of the topical agent, 1 hour after administration
Patient assessed health-related quality of life score | Up to 2 years postoperation
  This will be determined by a questionnaire/score
Difference in costs for hospital stay between using tranexamic acid and placebo | Duration of the hospital stay (an average of 2 weeks)
  Patient cost information will be gathered for the duration of the hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Ronald A Lehman, MD, Principal Investigator — Columbia University
Locations (4):
- United States (4):
  - University of California San Francisco Medical Center, San Francisco, California
  - Norton Leatherman Spine Center, Louisville, Kentucky
  - NYP/The Allen Hospital - CUIMC, New York, New York
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided